CLINICAL TRIAL: NCT04335474
Title: Surgical Versus Percutaneous Drainage in the Management of High Grade Pancreatic Trauma: A Prospective Controlled Study
Brief Title: Surgical Versus Percutaneous Drainage in the Management of High Grade Pancreatic Trauma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gao Tao, Dr, Nanjing PLA General Hospital
Other Study IDs: 2019NZKY-079-01
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Trauma; Pancreatic Trauma
Keywords: High-grade pancreatic trauma; Management strategy
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples analyses are performed by dedicated research centers: DNA, and RNA extraction for transcriptome analysis, histological analyzes, etc: The concentrations of cell-free DNA, cell-free nucleosomes, neutrophil elastase(NE) and myeloperoxidase (MPO) were measured in sera and plasma byHuman Cell Death Detection ELISA or sandwich ELISA. Pancreatic tissue was removed rapidly and divided into different parts for later analyses. One was used for confocal microscopy and one third was snap-frozen in liquid nitrogen for biochemical quantification of pancreatic myeloperoxidase (MPO), histone 3, and histone 4 levels, etc. One was fixed in formalin for histologic analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical drainage: Cases that have surgical management
  Interventions: Procedure: Surgical drainage strategy
- Percutaneous drainage: Cases that have the nonoperative management by percutaneous drainage
  Interventions: Procedure: Percutaneous drainage strategy

INTERVENTIONS:
Procedure: Surgical drainage strategy — A laparotomy is performed and the operative approach to pancreatic trauma can consist of laparotomy with drainage of the peripancreatic area, distal pancreatectomy with or without preservation of the spleen, Rouxen-Y pancreaticojejunostomy, and, more seldom, pancreaticoduodenectomy. The type of operation depends on the grade of the pancreatic lesion. Spleen-preserving surgery will be attempted to avoid the lifelong increased risk of infections after splenectomy. In case of trauma where multiple organs are involved and an acute laparotomy is performed, the damage control surgery must be applied and the pancreatic resection will be done as part of a staged surgery.
  Groups: Surgical drainage
Procedure: Percutaneous drainage strategy — The nonoperative management consists of close monitoring of the patient's clinical condition; repeated radiological investigations such as CT, ultrasound, and MRCP; monitoring of the amylase and lipase levels, initiation of post-pyloric enteral nutrition and parenteral nutrition. In addition, ERCP with the placement of a stent in the damaged pancreatic duct is used as part of the non-operative approach. Besides, percutaneous catheter drainage (PCD) management including ultrasound or CT-guided drainage of abdominal and peripancreatic fluid collections and pancreatic pseudocysts is applied to the HGPT patient.
  Groups: Percutaneous drainage

SUMMARY:
High-grade pancreatic injury is rare, and the reported complication and mortality are high.

The optimal management strategy according to high-grade injuries remains controversial.

The present study compares surgical drainage with percutaneous drainage in the management of High-grade pancreatic trauma.

DETAILED DESCRIPTION:
High-grade pancreatic trauma (HGPT), while uncommon, presents challenging diagnostic and therapeutic dilemmas to trauma surgeons. Multiple management strategies to HGPT have been reported, which was associated with a high level of morbidity and mortality rate. Besides, few prospective studies have investigated the optimal management strategy of patients with HGPT.

We aimed to compare surgical drainage with percutaneous drainage in the management of HGPT. To do so, the strategy is to integrate precise prospective clinical records extensive clinical treatment data in a large cohort of patients. All the clinical departments, participating in the study, include patients, with tight collaboration between Trauma, Intensive Care and Surgery departments. Demographics and clinical parameters are collected in a database.

Once after the diagnosis is confirmed, the inclusion of patients is performed, before scheduled hospital management, and after eligibility criteria checking, and consent form signature. During clinical management, several samples are collected: blood samples and surgical specimens. As a usual practice, post-operative treatment will be prescribed at the investigator's discretion, with the help of an acre-established algorithm. Several samples are also collected during this exam(blood and biological tissue sample).

At the same time as these managements, clinical data regarding medical history, pre-hospital treatment history, surgical history, treatment history, post-operative treatment if prescribed, treatment history between surgery and image logical diagnosis are recorded. Clinical data are also collected 12months after discharge during a scheduled visit organized as usual practice, for long-term study.

Several studies will be performed along with the cohort setting-up:

* Comparison of the diagnosis time and treatment time of patients with HGPT
* Study of surgical methods and intraoperative conditions in patients with HGPT
* Study of ICU resuscitation treatment of patients with HGPT
* Study of complication, ICU length of stay and hospital length of stay for patients with HGPT
* Study of nutritional support treatment for patients with HGPT
* Study of mortality and cost for patients with HGPT

All the biologic samples are stored on sites at -80°C, or at room temperature depending on the samples: Samples collected in tubes, are sent immediately, at room temperature, to the central pathology department in Jinling Hospital, Nanjing, China. All the other samples, stored at -80°C, are sent to the research institute of General Surgery, Medical School of Nanjing University, China.

Samples analyses are performed by dedicated research centers: DNA, and RNA extraction for transcriptome analysis, histological analyzes, etc:

Histological analyzes: Analysis of the structure of the excised pancreas or intestinal tissue.

Molecular Biology: Whole-genome expression analyses are performed using microarray and followed by Gene Ontology and clustering analyses.

Microbiota: Bacterial composition of the ileal mucosa-associated microbiota is analyzed at the time of surgery using 16S (MiSeq, Illumina) sequencing. The obtained sequences are analyzed using the Qiime pipeline to assess composition, alpha and beta diversity.

Immunology: Phenotype of immune cells: Immune cells are extracted from blood and fresh mucosal tissues. The phenotype of these cells is analyzed by cytometry.

Analysis of neutrophil extracellular traps:

The concentrations of cell-free DNA, cell-free nucleosomes, neutrophil elastase(NE) and myeloperoxidase (MPO) were measured in sera and plasma byHuman Cell Death Detection ELISA or sandwich ELISA.

Pancreatic tissue was removed rapidly and divided into different parts for later analyses. One was used for confocal microscopy and one third was snap-frozen in liquid nitrogen for biochemical quantification of pancreatic myeloperoxidase(MPO), histone 3, and histone 4 levels, etc. One was fixed in formalin for histologic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with high-grade pancreatic trauma by surgery
* Patient diagnosed with high-grade pancreatic trauma by computed tomography
* Patient diagnosed with high-grade pancreatic trauma by Endoscopic retrograde cholangiopancreatography (ERCP)
* Patient diagnosed with high-grade pancreatic trauma by Magnetic resonance cholangiopancreatography (MRCP)

Exclusion Criteria:

* The patient underwent chemotherapies or radiotherapy
* Immune system disease
* Low-grade pancreatic trauma
* Accompanied by severe trauma to other organs
* End-stage chronic organ failure
* With multiple severe injuries
* Died within 24 h of admission
* Younger than 18 years
* Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who treated for High-grade pancreatic injuries at a national Level 1 trauma center
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  All cause mortality within 28 days

SECONDARY OUTCOMES:
Pancreatic associated complications | Through study completion, an average of 1 year
  Complications due to pancreatic problems
Non-pancreatic associated complications | Through study completion, an average of 1 year
  Abdominal complications of non-pancreatic problems
Organ failure | 28 days
  Organ failure caused by organ dysfunction
Systematic complication | 28 days
  Complications such as pneumonia, abdominal sepsis, etc
Days on total parenteral nutrition | Through study completion, an average of 6 months]
  Treatment time of parenteral nutrition support required during hospitalization
Time to enteral nutrition | Through study completion, an average of 6 months
  Time from management to initiate enteral nutrition in pancreatic injury patients
Days to clear liquids | Through study completion, an average of 6 months
  The time when the drainage tube is pulled out after the patient's abdominal liquids cleated
Days to regular diet | Through study completion, an average of 6 months
  The time from the treatment to the normal eating of patients with pancreatic trauma
Postoperative 28-day adverse effects | 28 days
  All cause adverse effects within 28 days
Hospital length of stay | Through study completion, an average of 6 months
  Length of hospital stay
Intensive Care Unit length of stay | Through study completion, an average of 6 months
  Length of Intensive Care Unit stay

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei Ding, MD, Study Director — Medical School of Nanjing University
Locations (1):
- Jinling Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: No